CLINICAL TRIAL: NCT06663774
Title: Development of a Judo Specific Reactive Agility Test: a Reliability and Validity Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Turgut, PT, PhD, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GO 21/1091
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-01

CONDITIONS: Validation Study; Athletic Performance
Keywords: Reactive; Agility; Performance; Reliability; Validity; Judo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Judokas (Experimental): Judokas between the age of 18-45 with at least 3 years of judo experience who are actively doing judo training minimum of 300 minutes in a weak.
  Interventions: Diagnostic Test: Physical Fitness Tests

INTERVENTIONS:
Diagnostic Test: Physical Fitness Tests — Ippon Reactive Agility Test (IRAT), Y-Balance Test, Upper-Quarter Y Balance Test, Flamingo Balance Test, Flamingo Balance Test, Standing Long Jump Test, 20m Sprint Test, Hand Grip Test, T-Agility Test, Nelson Hand Reaction Test, Judo Specific Fitness Test

SUMMARY:
Primary aim of this study is to develop a new reactive agility test spesific for Judokas and evaluate it's validity and reliability. Secondary aim is the investigation of relationship between reactive agility performance score and some of the physical fitness parameter scores related to health and performance.

ELIGIBILITY:
Inclusion Criteria:

* Active judo training of minimum 300 minutes in a week.
* At least 3 years of Judo experiance
* No acute injury or illness that prevents judo training
* No use of drug or medicine that can/may affect noromusculer control

Exclusion Criteria:

* Major trauma in 6 months prior to study
* Judokas that can't complete the test properly

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Validity and reliability | 3-5 days
  pearson's correlation 2 tailed analysis; >0,60 good, 0,31-0,59 medium, <0,30 bad

SECONDARY OUTCOMES:
Relationship between the IRAT and other physical fitness parameters | 3-5 days
  Pearson correlation coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided